CLINICAL TRIAL: NCT06662084
Title: Impact of Temporary Mechanical Circulatory Support (tMCS) on Cytochromes P450 Activity Measured with Dried Blood Spot
Brief Title: The ECMOCYP (cytochromes P450 Activity) Study
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: Jean Terrier (Unknown); Benjamin Assouline (Unknown); Raphël Giraud (Unknown); Karim Bendjelid (Unknown); Caroline Samer (Unknown); Youssef Daali (Unknown); Anastasia Zaslavskaya (Unknown)
Responsible Party: Principal Investigator, Jean Terrier, MD, PharmD, PhD, University Hospital, Geneva
Other Study IDs: 2023-01398
Record Dates: First submitted 2024-09-13; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: ECMO; Cardiogenic Shock; Temporary Mechanical Circulatory Support
Keywords: ecmo; cardiogenic shock; Temporary Mechanical Circulatory Support; TMCS; CYP450; phenotyping; genotyping
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Phenotype

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Temporary mechanical circulatory support group: Male and female patients presenting a refractory cardiogenic shock, requiring temporary mechanical circulatory support (tMCS), with either the use of veno-arterial extracorporeal membrane oxygenation (VA-ECMO) or a micro-axial pump device (Impella® CP).
  Interventions: Diagnostic Test: phenotype
- Control group: Male and female patients in cardiogenic shock according to the SCAI (Society for Cardiovascular Angiography and Interventions) ESC (European Society of Cardiology) definition and not requiring or not eligible to temporary mechanical circulatory support (tMCS). (e.g. ECMO, Impella®, intra-aortic balloon pump)
  Interventions: Diagnostic Test: phenotype

INTERVENTIONS:
Diagnostic Test: phenotype — Eligible patients will receive orally the cocktail probe drugs ( via a naso-gastric tube at D3 after tMCS implantation or after the beginning of the cardiogenic shock for the control group) and via an oral administration at 14 days after tMCS explantation (or cardiogenic shock termination for the control group defined as: no need to use inortropic or vasopressive agent and absence of organ insufficiency). The phenotyping probe drugs of the Geneva Cocktail will be given as: one capsule containing the remaining probe 'cocktail' drugs. According to clinical experience in our intensive care unit department, inflammation related to tMCS peaks at D3 after tMCS implantation.
  Blood samples will be collected from the central venous line 2 hours after drug administration for CYP phenotyping and genotyping. Inflammatory markers blood levels (Il-6, TNF-α, Il-1β, IFN-γ) will be measured at tMCS implantation or shock initiation and at the same time than CYP phenotyping.
  Other Names: CRP; IL-6; TNF-alpha; IL-1β; IFN-γ

SUMMARY:
Prospective open label observational study including patients requiring a tMCS (VA-ECMO or Impella® CP) or in in cardiogenic shock according to the SCAI (Society for Cardiovascular Angiography and Interventions) ESC (European Society of Cardiology) definition 41,42 and not requiring or not eligible to tMCS (ECMO, Impella®, intra-aortic balloon pump) (control group).

DETAILED DESCRIPTION:
The Geneva cocktail will be administered on 2 occasions at D3 after tMCS implantation (or start of the cardiogenic shock) and 14 days after tMCS explantation (or cardiogenic shock termination defined as: no need to use inortropic or vasopressive agent and absence of organ insufficiency)

Primary endpoint:

* Evaluate the impact of tMCS on the activity of CYPs as measured with metabolic ratios MRs (CYP activity at
* D3 post tMCS implantation and 14 days after tMCS explantation vs the activity of CYPs in the control group.

Secondary endpoints:

* Evaluate the correlation between the activity of CYPs and IL-6 levels
* Evaluate the correlation between the activity of CYPs and CRP levels
* Evaluate the correlation between the activity of CYPs and TNF-α levels
* Evaluate the correlation between the activity of CYPs and IL-1β levels
* Evaluate the correlation between the activity of CYPs and IFN-γ levels
* Compare CYP activity vs expected CYP activity based on patients' CYP genotyping
* Compare CYP activity between VA-EMCO and micro-axial pump device (Impella® CP)

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients presenting a refractory cardiogenic shock, requiring temporary mechanical circulatory support (tMCS), with either the use of veno-arterial extracorporeal membrane oxygenation (VA-ECMO) or a micro-axial pump device (Impella® CP).
* Male and female patients in cardiogenic shock according to the SCAI (Society for Cardiovascular Angiography and Interventions) ESC (European Society of Cardiology) definition and not requiring or not eligible to temporary mechanical circulatory support (tMCS). (e.g. ECMO, Impella®, intra-aortic balloon pump) (control group)
* Age > 18 years old
* Comprehension of French
* Ability to give consent (consent will be sought from the therapeutic representative or from relatives as the patient will be sedated and intubated. Definitive consent will be sought at patient's second blood sample planned after tMCS explantation (in case of patient's favorable outcome).

Exclusion Criteria:

* Male and female patients presenting a refractory ARDS requiring veno-venous extracorporeal membrane oxygenation (VV-ECMO)
* Inability to receive the Geneva cocktail by enteral way
* Severe or terminal Renal impairment (defined as GFR<30ml/min according to Cockroft-Gault)
* Severe chronic hepatic insufficiency (CHILD B-C)
* Sensitivity to any of the drugs used in the Geneva Cocktail
* Intake of drugs altering CYPs activity (Strong inhibitor or inducer based on https://www.hug.ch/sites/hde/files/structures/pharmacologie_et_toxicologie_cliniques/a5_cytochromes_6_2.pdf)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Male and female patients presenting a refractory cardiogenic shock, requiring temporary mechanical circulatory support (tMCS), with either the use of veno-arterial extracorporeal membrane oxygenation (VA-ECMO) or a micro-axial pump device (Impella® CP).
  * Male and female patients in cardiogenic shock according to the SCAI (Society for Cardiovascular Angiography and Interventions) ESC (European Society of Cardiology) definition and not requiring or not eligible to temporary mechanical circulatory support (tMCS). (e.g. ECMO, Impella®, intra-aortic balloon pump) Hospitalised in intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of temporary mechanical circulatory support on the activity of CYPs as measured with metabolic ratios MRs (CYP activity at D3 post tMCS implantation and 14 days after tMCS explantation vs the activity of CYPs in the control grou | During the ECMO
  CYP450 3A4, 2C19, 2D6, 2B6, 1A2 activity will be assessed in using the metabolic ratio of the following probe respectively: midazolam, esomeprazole, dextrometorphan, bupropion and caffein.

SECONDARY OUTCOMES:
Evaluate the correlation between the activity of CYPs and IL-6 levels | During the ECMO
Evaluate the correlation between the activity of CYPs (MRs) and CRP levels | During the ECMO
Evaluate the correlation between the activity of CYPs (MRs) and TNF-α levels | During the ECMO
Evaluate the correlation between the activity of CYPs (MRs) and IL-1β levels | During the ECMO
Evaluate the correlation between the activity of CYPs (MRs) and IFN-γ levels | During the ECMO
Compare CYP activity vs expected CYP activity based on patients' CYP genotyping | During the ECMO
  CYP phenotyping based classification in metabolizer status (UM, NM, IM or PM) using metabolic ratios will be compared to genotyping based classification from the star allele nomenclature according to Pharmacogene Variation (PharmVar) Consortium. ).
Compare CYP activity based on phenotyping between VA-EMCO and micro-axial pump device (Impella® CP) | During the ECMO
  CYP450 CYP3A4, 2C19, 2D6, 2C19, 1A2 activity will be determined as mentionned for the primary issue and will be compared between the groups VA-ECMO and micro-axial pump device

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided